CLINICAL TRIAL: NCT01479816
Title: Urinary Continence Index for Prediction of Urinary Incontinence in Older Women
Status: Completed | Type: Observational
Sponsor: Ananias Diokno (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Ananias Diokno, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: E2011-047; 1R01AG038673 (NIH)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Urinary Incontinence
Keywords: continence; index
MeSH Terms: conditions — Urinary Incontinence; Erythema Multiforme

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will analyse existing data to establish a clinically useful index to predict those women who are more likely to become incontinent. This would create significant opportunities for focused prevention and early intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Women

Exclusion Criteria:

* Men

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 55 years and older
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Index Estimation for Urinary Incontinence Prediction | 2 years
  Several risk factors identified can serve as an index in predicting the development of urinary incontinence in elderly women.

SECONDARY OUTCOMES:
Predictive Reliability of Urinary Incontinence Index and its Validation | 3 years
  The urinary continence index developed in Outcome measure 1 will reliably predict the development of urinary incontinence in women when tested against existing datasets.

CONTACTS AND LOCATIONS:
Overall Officials: Ananias Diokno, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Oakland University, Rochester, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No